CLINICAL TRIAL: NCT00109187
Title: Open-Label Extension Study II of Xolair (Omalizumab) in Moderate to Severe, Persistent Asthma Subjects Who Completed Study Q2143g (ALTO)
Brief Title: An Extension Study of Xolair in Moderate to Severe, Persistent Asthma Patients Who Completed Study Q2143g
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Masking: None | Purpose: Treatment
Other Study IDs: Q2461g
Record Dates: First submitted 2005-04-26; First posted 2005-04-26 (Estimated); Last update posted 2013-06-21 (Estimated); Status verified 2013-06

CONDITIONS: Asthma
Keywords: Moderate Persistent Asthma; Severe Persistent Asthma
MeSH Terms: conditions — Asthma | interventions — Omalizumab

INTERVENTIONS:
Drug: Xolair (omalizumab)

SUMMARY:
This is a Phase IIIb, multicenter, open-label, extension study available to subjects who successfully complete Study Q2143g and have not participated in Study Q2195g. Subjects should be registered via the IVRS (Interactive Voice Response System) within 48 hours prior to their baseline visit. All subjects in this study will be treated with Xolair for 24 weeks. Subjects in the New Treatment Group may require additional visits for study drug injections (as frequently as every 2 weeks). Data collection during these additional visits will be limited to the assessment of adverse events. The study will evaluate all serious and nonserious adverse events, laboratory assessments, data on asthma exacerbations, and concomitant medication usage.

ELIGIBILITY:
Inclusion Criteria:

* Successful completion of the 24-week study period in Study Q2143g
* Signed informed consent (in the case of a minor, consent must be given by the child's parent or legally authorized representative)
* For subjects who have never received Xolair, a serum IgE level >=30 IU/mL and <=1300 IU/mL and have a body weight >=20 kg and <=150 kg
* Females of childbearing potential must, in the opinion of the investigator, be using an effective method of contraception to prevent pregnancy and agree to continue to practice an acceptable method of contraception for the duration of their participation in the study.

Exclusion Criteria:

* Thrombocytopenia as evidenced by a platelet count of <100,000/uL
* Pregnant or breastfeeding
* Significant systemic disease (e.g., infection, hematologic, renal, hepatic, coronary heart disease or other cardiovascular diseases, endocrine or gastrointestinal disease) within the previous 3 months
* History of neoplasia
* Any systemic condition requiring regular administration of an immunoglobulin
* Known hypersensitivity to any ingredients of Xolair, including excipients (sucrose, histidine, polysorbate 20)
* History of noncompliance with medical regimens
* Current participation in a study using an investigational new drug other than Xolair
* Participation in Study Q2195g

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0
Dates: Start 2002-06; Study Completion 2003-04 (Actual)